CLINICAL TRIAL: NCT05261282
Title: Mindful Hand Hygiene to Reduce Infections Among Veterans While Enhancing Provider Well-Being
Brief Title: Mindful Hand Hygiene for Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-097
Record Dates: First submitted 2022-02-04; First posted 2022-03-02 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Burnout; Mental Health
Keywords: Mindfulness; Hand Hygiene; Health Personnel
MeSH Terms: conditions — Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a multi-center, repeat-measures, randomized controlled mixed-methods trial. At each study site the participating physician teams and nursing units will be randomly assigned into one of two study arms (intervention/control). For physician teams, this will occur on a rolling basis for 12 months with 2 physician teams randomly selected at each site each month for participation (1 intervention, 1 control). For nurses, 2-4 hospital units at each study site will be assigned to either intervention or control for the study period.
Who Masked: Outcomes Assessor
Masking Description: The research staff who conduct the hand hygiene observations for the physician teams will not know the randomization status of the physician teams. The investigators are unable to mask the research assistants from the randomization status of the nursing units.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindful Hand Hygiene Intervention (Experimental): Participants in the Mindful Hand Hygiene Intervention will complete the same surveys as participants in the Control Arm at baseline, post-intervention, and 6-months post-intervention. Data will also be collected on baseline hand-hygiene rates during the habituation period, intervention period, and 3-12 months post-intervention. In addition, intervention participants will be asked to complete 3 mindfulness online educational modules and attend group-facilitated discussions on mindfulness. They will be offered the option of using a mobile application program "Mindfulness Coach" to enhance their mindfulness practices. A key message of the intervention is using hand hygiene as a prompt to practice mindfulness.
  Interventions: Behavioral: Mindful Hand Hygiene
- Control Arm (No Intervention): Participants that are assigned to the control arm will be observed for hand hygiene adherence and duration during the habituation period, intervention period, and 3-12 months post-intervention. They will also be asked to complete study surveys at baseline, post-intervention and 6-months post intervention. They will not receive any of the intervention components.

INTERVENTIONS:
Behavioral: Mindful Hand Hygiene — Physicians and nurses randomized to the intervention arm will receive mindfulness education and tools to prompt mindfulness during hand hygiene.
  Arms: Mindful Hand Hygiene Intervention

SUMMARY:
The purpose of this study is to test an intervention focused towards promoting mindfulness among VA physicians and nurses. Mindfulness is a tool that can help people focus. It helps clear the mind of distractions and biases. Some physicians and nurses will be randomized to receive the study intervention, while others will not. The study intervention will include the following: 1) education about mindfulness; 2) group discussions about mindfulness; and 3) an optional mobile app to promote mindfulness. Participants randomized to the intervention will be encouraged to use the act of cleansing their hands as a prompt for practicing mindfulness. The study will test if this intervention will increase physician and nurse mindfulness. It will also test if it leads to improved well-being and use of proper hand hygiene.

DETAILED DESCRIPTION:
Physician and nurse well-being is important for providing high quality patient care. Many physicians and nurses suffer from stress, fatigue, psychological distress, depression, and burnout. This can lead to poor patient care. In this study, the investigators will use a repeat-measures randomized controlled mixed-methods trial to evaluate an intervention designed to improve healthcare provider well-being. The intervention will help physicians and nurses practice moments of mindfulness. Mindfulness is paying attention to the present moment. It can help people feel more aware instead of feeling like they are running on automatic pilot. The investigators will test if practicing mindfulness while cleaning hands before and after seeing patients will lead to improved well-being and hand hygiene.

This is a multi-center, repeat-measures randomized controlled mixed-methods trial that will last 3 years. The primary objective of this phase 1/2 clinical trial is to implement and evaluate an intervention to improve physician & nurse well-being through promoting mindfulness. Secondary objectives include monitoring physician and nurse hand hygiene adherence and duration and conducting a qualitative assessment to evaluate the intervention. The study will enroll approximately 334 physicians and nurses from 2 VA Medical Centers (LTC Charles S. Kettles VA Medical Center, Ann Arbor, MI; and Michael E. DeBakey VA Medical Center, Houston, TX).

The proposed study will focus on Internal Medicine physicians who are part of inpatient care teams and nurses providing care on medical and medical/surgical units at LTC Charles S. Kettles VAMC in Ann Arbor, MI and MEDVAMC in Houston, TX. Medical students, surgical physicians, and physicians on sub-specialty teams will not be included. At both participating facilities the inpatient care teams are predominately composed of 1 attending, 1 senior resident, 2 interns, and up to 3 medical or physician assistant students. Interns and senior residents are usually assigned to a team for 4-week blocks (occasionally 2 weeks), while attendings rotate approximately every 2 weeks. The Ann Arbor VAMC has 3 medical or medical/surgical inpatient units, while MEDVAMC has 5 units. At both facilities each nursing unit employs between 20-30 nurses. The investigators will aim to recruit approximately 30 attendings, 72 residents and 40 nurses at Ann Arbor VAMC. As MEDVAMC is larger, with a greater number of inpatient care teams and nursing units than the Ann Arbor VAMC, the investigators will aim to recruit approximately 40 attendings, 72 residents and 80 nurses. The target study sample size is a total of 334 physicians and nurses (167 intervention/167 control). For Aim 3, the investigators plan to interview approximately 8 physician team members and 4-6 nurses from the intervention arm at each site.

Randomization: At each study site the participating physician teams and nursing units will be randomly assigned into one of two study arms (intervention/control). For physician teams, this will occur on a rolling basis for 12 months with 2 physician teams randomly selected at each site each month for participation (1 intervention, 1 control). Once randomized, an email will be sent to the initial attending of the team introducing the study and seeking approval for their team to participate in the randomized controlled trial. If the attending physician from a team refuses participation, the next team identified from the randomized list will be approached to participate. If a new attending joins the team mid-month, they will be approached to participate in the study, but will be automatically assigned to the same randomization group as the rest of their team.

Similarly, a total of 2 medical/surgical units from the Ann Arbor VA (1 intervention, 1 control) and 4 medical/surgical units from Houston VA (2 intervention, 2 control) will be randomly selected to participate in the nurse portion of the project. The nurse manager for each selected unit will then be approached to obtain approval for the unit to participate. If a nurse manager declines, the next unit on the list will be selected.

An independent statistician will allocate the physician teams and nursing units at both study sites in a concealed fashion, using a computer-generated randomization schema. The physicians and nurses from the intervention groups will receive both independent and group-facilitated mindfulness education, will be encouraged to use a mindfulness mobile app as a practice reminder and additional resource, and instructed to integrate moments of mindfulness with repeated episodes of hand hygiene during the course of caring for patients. The control groups will receive no such education or intervention and will continue providing care as usual.

Recruitment and Control Arm: Potential subjects will be recruited via email or in-person communications. Everyone who consents to participate (regardless of study arm) will be asked to complete baseline surveys containing validated scales measuring dispositional mindfulness, well-being, and hand hygiene perceptions. The Five Facet Mindfulness Questionnaire (FFMQ) is a validated instrument with favorable psychometric properties and consists of 39 questions. Additionally, participants will be asked to complete the Well-Being Index (WBI). The 9-question WBI assesses distress across a variety of dimensions including fatigue, depression, burnout, stress, and quality of life, and has been validated for use in physicians, residents, and nurses. Participants will also be asked to complete 8 questions on healthcare-associated infections and hand hygiene perceptions selected from the Perceptions Survey for Healthcare Workers (PSHW) developed by the World Health Organization. Similar to other studies on hand hygiene perceptions guided by the constructs based on the Theory of Planned Behavior, the selected PSHW questions cover behavioral, normative, and control beliefs, as well as self-reported hand hygiene adherence. Participants will also be asked whether they meditate or perform any form of internal reflection prior to the study, as this may influence performance during the intervention. Completing the full survey questionnaire will take approximately 10 minutes.

Habituation Period: To collect baseline data on hand hygiene adherence and duration for both study arms and to habituate providers to the presence of observers, 1 month of covert, unit-based hand hygiene observations will be conducted. Observation of hand hygiene adherence will include hand hygiene prior to patient room entry and after exiting the patient room. Hand hygiene observers will not enter patient rooms or interfere in patient care. Observation of hand hygiene duration will be done when providers exit patient rooms, as observing hand hygiene duration upon room entry will not be feasible since observers will not enter patient rooms and providers may practice hand hygiene while entering the patient room.

Intervention Activities: Participants in the intervention will be asked to complete 3 self-directed online education modules on mindful practice developed by the Ohio State University Mind-Body Skills Training for Resilience, Effectiveness, and Mindfulness (STREAM) program (http://mind-bodyhealth.osu.edu). Subjects will receive compensation for completion of each online training module completed outside of their working hours. Participants will also be asked to participate in group-facilitated discussions with their site mindfulness champion where they will discuss using mindfulness during their work day. During these discussions, participants will be instructed to use the act of hand hygiene as a moment to pause and reflect - a mindful moment. The guided discussions will be recorded, transcribed, and used in the qualitative evaluation of the intervention. Intervention participants will also be given the option of using a self-directed mobile application to enhance their mindfulness education and practice. The study will use the Mindfulness Coach mobile app, which was developed by researchers at the National Center for Posttraumatic Stress Disorder, Dissemination & Training Division at the VA Palo Alto Health Care System.

Post-Intervention Activities: The same measures that were collected during the pre-intervention period will again be collected during the post-intervention period. Subjects will be asked to complete the same survey once the 1-month intervention has ended. They will also be asked to complete the survey again 6-months post-intervention to assess sustainability. The research assistants will again conduct covert direct observations of hand hygiene moments during the intervention phase and 3-12 months post-intervention. Select subjects will also be asked to participate in qualitative interviews after the intervention is complete to provide: views on the intervention; overall perceptions of and experiences with mindfulness; barriers encountered while trying to implement the intervention during clinical practice; personal sense of well-being and whether or not the intervention had any effect on well-being; perceptions on whether or not practicing mindfulness during hand hygiene had any impact on hand hygiene adherence; and the potential benefits of using mindfulness in the clinical setting.

Data Analysis: Differences in hand hygiene adherence and duration between intervention and control groups will be assessed using Fisher's exact test and t-test, as appropriate. Risk differences in adherence to duration of hand hygiene will be calculated for both intervention and control groups. Because the primary outcomes for Aim 1 (i.e., hand hygiene adherence and duration) are expected to occur frequently, the investigators will use generalized linear models to evaluate differences in hand hygiene adherence and duration for the intervention versus control group, with the Poisson distribution (log link) and robust error variance. Models will account for provider type and level, and will incorporate clustering by physician team (and separately for nursing unit). Statistical significance will be calculated for the intervention (intervention vs. control) coefficient.

As a secondary outcome for Aim 1, the investigators will assess changes and differences in hand hygiene perception based on responses to select questions from the PSHW. For Aim 2, mindfulness will be based on responses to the FFMQ and well-being will be based on responses to the WBI. Survey scales will be scored according to the published algorithms. Descriptive statistics will be used to summarize participant scores from pre- and post-intervention, as well as 6-month post-intervention follow-up assessments. Within-group paired-samples t-tests will be used to test for improvement in participant scores across the baseline, post-intervention (~14 days for physicians and 1-month for nurses), and 6-month post-intervention follow-up periods, for the intervention and control groups separately. Analyses will use list-wise deletion for missing data. Participants not completing all surveys will still be included in any analysis for which they provide data. For all analyses, p-values less than 0.05 will be considered significant and all tests will be two-tailed. Analysis of covariance (ANCOVA) models will then be used to assess relative changes in mindfulness, well-being, and hand hygiene perceptions across groups, the most direct test of discriminant validity. In these models, post-test scores will be predicted by group status controlling for pre-test scores.

ELIGIBILITY:
Inclusion Criteria:

* Nurses on participating unit
* Physician on an inpatient medical team, including attending, senior resident, and intern physicians

Exclusion Criteria:

* Medical students
* Surgical attendings
* Physicians on sub-specialty teams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
The Five Facet Mindfulness Questionnaire (FFMQ) - Baseline | Month 0
  The Five Facet Mindfulness Questionnaire (FFMQ) is a validated instrument with favorable psychometric properties and consists of 39 questions. Scores are combined into the following subscales - Observing, Describing, Acting with Awareness, Nonjudging, Nonreactivity as well as a total score. Scores on the Observing, Describing, Acting with Awareness, and Nonjudging subscales range from 8-40, while the Nonreactivity subscale ranges from 7-35. The total FFMQ scores can range from 39-195. Lower scores mean less mindful, while higher scores indicate the respondent is more mindful. Scores can also be averaged for each subscale (1-5)
Perceptions Survey for Healthcare Workers (PSHW) - Baseline | Month 0
  Participants will also be asked to complete 8 questions on healthcare-associated infection and hand hygiene perceptions selected from the Perceptions Survey for Healthcare Workers (PSHW) developed by the World Health Organization. PSHW questions cover behavioral, normative, and control beliefs, as well as self-reported hand hygiene adherence. Individual question responses will be assessed on scales of 1-4, 1-7 or 0-100. Higher scores indicate higher importance of the practice.
Well-Being Index - Baseline | Month 0
  The 9-question WBI assesses distress across a variety of dimensions including fatigue, depression, burnout, stress, and quality of life, and has been validated for use in physicians, residents, and nurses. Scores range from -2 (low-risk) to 9 (high risk).
The Five Facet Mindfulness Questionnaire (FFMQ) - Post-Intervention | Month 1
  The Five Facet Mindfulness Questionnaire (FFMQ) is a validated instrument with favorable psychometric properties and consists of 39 questions. Scores are combined into the following subscales - Observing, Describing, Acting with Awareness, Nonjudging, Nonreactivity as well as a total score. Scores on the Observing, Describing, Acting with Awareness, and Nonjudging subscales range from 8-40, while the Nonreactivity subscale ranges from 7-35. The total FFMQ scores can range from 39-195. Lower scores mean less mindful, while higher scores indicate the respondent is more mindful. Scores can also be averaged for each subscale (1-5).
Well-Being Index - Post-Intervention | Month 1
  The 9-question WBI assesses distress across a variety of dimensions including fatigue, depression, burnout, stress, and quality of life, and has been validated for use in physicians, residents, and nurses. Scores range from -2 (low-risk) to 9 (high risk).
Perceptions Survey for Healthcare Workers (PSHW) - Post-Intervention | Month 1
  Participants will also be asked to complete 8 questions on healthcare-associated infection and hand hygiene perceptions selected from the Perceptions Survey for Healthcare Workers (PSHW) developed by the World Health Organization. PSHW questions cover behavioral, normative, and control beliefs, as well as self-reported hand hygiene adherence. Individual question responses will be assessed on scales of 1-4, 1-7 or 0-100. Higher scores indicate higher importance of the practice.
The Five Facet Mindfulness Questionnaire (FFMQ) - 6-months Post-Intervention | Month 7
  The Five Facet Mindfulness Questionnaire (FFMQ) is a validated instrument with favorable psychometric properties and consists of 39 questions. Scores are combined into the following subscales - Observing, Describing, Acting with Awareness, Nonjudging, Nonreactivity as well as a total score. Scores on the Observing, Describing, Acting with Awareness, and Nonjudging subscales range from 8-40, while the Nonreactivity subscale ranges from 7-35. The total FFMQ scores can range from 39-195. Lower scores mean less mindful, while higher scores indicate the respondent is more mindful. Scores can also be averaged for each subscale (1-5).
Well-Being Index - 6-months Post-Intervention | Month 7
  The 9-question WBI assesses distress across a variety of dimensions including fatigue, depression, burnout, stress, and quality of life, and has been validated for use in physicians, residents, and nurses. Scores range from -2 (low-risk) to 9 (high risk).
Perceptions Survey for Healthcare Workers (PSHW) - 6-months Post-Intervention | Month 7
  Participants will also be asked to complete 8 questions on healthcare-associated infection and hand hygiene perceptions selected from the Perceptions Survey for Healthcare Workers (PSHW) developed by the World Health Organization. PSHW questions cover behavioral, normative, and control beliefs, as well as self-reported hand hygiene adherence. Individual question responses will be assessed on scales of 1-4, 1-7 or 0-100. Higher scores indicate higher importance of the practice.

SECONDARY OUTCOMES:
Hand Hygiene - Habituation | Month 0
  Research assistants will conduct covert direct observations of hand hygiene moments during weekdays. The metric will include whether the physician or nurse used hand rub, washed with soap and water, or did not wash their hands before entering and after exiting a patient room. Duration of hand hygiene will also be measured upon room exit.
Hand Hygiene - Intervention | Month 1
  Research assistants will conduct covert direct observations of hand hygiene moments during weekdays. The metric will include whether the physician or nurse used hand rub, washed with soap and water, or did not wash their hands before entering and after exiting a patient room. Duration of hand hygiene will also be measured upon room exit.
Hand Hygiene - Post-Intervention | Months 2-13
  Research assistants will conduct covert direct observations of hand hygiene moments during weekdays. The metric will include whether the physician or nurse used hand rub, washed with soap and water, or did not wash their hands before entering and after exiting a patient room. Duration of hand hygiene will also be measured upon room exit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Todd Greene, PhD MPH BS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Sanjay K. Saint, MD MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created. Members of the scientific community who would like a copy of the final data sets (i.e., data sets underlying any publication) from this study can request a copy by e-mailing Jennifer Burns at Jennifer.Burns@va.gov. They should state their reason for requesting the data and their plans for analyzing the data. Final data sets will be copied onto a DVD. Limited data sets will be encrypted; and the password will be sent to the requestor via e-mail. The DVD will be sent to the requestor via FedEx.
Supporting Information: SAP
Time Frame: After the final publication from this study.
Access Criteria: De-identified data will be provided after requesters sign a Letter of Agreement (LOA) detailing the mechanisms by which the data will be kept secure. The LOA will also state that the recipient will not attempt to identify any individual in the data, will not share the data outside of their research team, and will provide information on any files to be linked to the data. The dataset will not include PII and all dates will be changed to integers to allow for calculation of time periods.

REFERENCES:
- [Result] Kirykowicz K, Jaworski B, Owen J, Kirschbaum C, Seedat S, van den Heuvel LL. Feasibility, acceptability and preliminary efficacy of a mental health self-management app in clinicians working during the COVID-19 pandemic: A pilot randomised controlled trial. Psychiatry Res. 2023 Nov;329:115493. doi: 10.1016/j.psychres.2023.115493. Epub 2023 Sep 24. PMID 37778231

DOCUMENTS (1):
  • Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT05261282/ICF_000.pdf